CLINICAL TRIAL: NCT06041347
Title: Evaluation of the Learning Curve for the Visualization of Sacral Nerve Roots and Sacral Plexus on Gynecological Transvaginal Ultrasound - PlexUS Study
Brief Title: Learning Curve for the Visualization of Sacral Plexus on TVS
Acronym: PlexUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Semmelweis University (Other)
Collaborators: Jagiellonian University (Other); Charles University, Czech Republic (Other); St John of God Hospital, Vienna (Other)
Responsible Party: Sponsor
Other Study IDs: Semmelweis University Szabó G
Record Dates: First submitted 2023-09-05; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Endometriosis; Nerve Sheath Tumor; Radiculopathy
MeSH Terms: conditions — Endometriosis; Nerve Sheath Neoplasms; Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasound — Preoperative detection with TVUS of proximity or the involvement of the sacral nerve roots in women diagnosed with deep endometriosis or other benign or malignant pelvic tumors would also contribute to the safety of surgical interventions (e.g laparoscopy, tru-cut biopsy) It aslo provides correct counseling and select the appropriate surgical team and assess the likely operative complexity of the surgery. Until now the diagnosis was based on MRI.

SUMMARY:
The purpose of this prospective study was to evaluate the learning curve of TVUS (transvaginal ultrasound) for the visualization of sacral nerve roots and sacral plexus on gynecological transvaginal ultrasound. The investigators aim to evaluate to evaluate the number needed to gain competence or to review the level of competence.

DETAILED DESCRIPTION:
For each patient, the fellows are blinded to the clinical and surgical history. The investigators will be aware that all patients were being evaluated for pelvic pain or endometriosis. The expert sonographer assess the patient and visualized the sacral roots and the sacral plexus first as part of the advanced TVUS examination for endometriosis.

TVUS examination will conducted in six steps eas follows in six successive steps. All women will be asked to empty their bladder prior to examination. TVUS scans will be performed in the lithotomy position in a standardized fashion using a transvaginal probe Step 1: First the probe will inserted into the anterior vaginal fornix. The uterus is examined in the midsagittal view on the longitudinal section to identify the cervix and the uterine cavity. The image is frozen with time displayed on the screen, which was marked as Time 1.

Step 2: The image is unfrozen and at the level of the inner cervical meatus the transducer is rotated 90 degrees counterclockwise to obtain a transverse scan.

Step 3: Then the probe is immediately moved towards the right lateral fornix pointing towards the uterine vessels, which appear as hypoechoic bands. Behind these structures, a thick hyperechoic band - the left uterosacral ligament -appears, starting from the cervix and pointing laterally in a semi horizontal direction. By rotating the probe the uterosacral ligament is then followed from medial to lateral, up to the lateral pelvic wall. The obturator internus muscle covers most of the lateral wall of the pelvis minor, which - in transverse scan - is a hypoechoic thin band just lateral to the uterosacral ligament. On the lateral side of the muscle a continuous bright white band is seen, corresponding to the body of the ischium.

Step 4: Sweeping the probe medially and pushing it superior the hypoechoic obturator internus muscle and the hyperechoic ischium are followed ending at the greater sciatic foramen. At this point transverse and oblique sections of the branches of the anterior division of the internal iliac vessels became visible. Deeper to the vessels the hypoechoic muscle fiber bundles with intervening echogenic perimysium, the piriformis muscle, and a bright white line, the anterior surface of the sacrum are visualized. Between the vessels and the piriformis muscle on conventional gray scale B mode the sacral roots of the sacral plexus (SP) appear in longitudinal section, with a typical "bundle of straw" appearance: hypoechoic bands, with echogenic septae. The hypoechoic areas correspond to nerve fascicles, while the hyperechoic septae correspond to the inner and outer epineurium. In transverse section, the nerves have a "honeycomb" shape echotexture.

Step 5: Pushing the transducer superior color Doppler and pulse wave Doppler can be used to differentiate blood vessels from the ureter on the lateral pelvic wall and to identify the branching of the internal iliac artery. From the posterior division rises the superior gluteal artery and from the anterior division originates the inferior gluteal artery. Both of them exiting the pelvis between the ischium and the sacrum. The former runs between the lumbosacral trunk and the ventral ramus of the S1 nerve and leaves the pelvis superior to the piriformis muscle. The inferior gluteal artery passes usually posteriorly between S2 and S3 roots, and leaves the pelvis together with the sciatic nerve, inferior to the piriformis muscle near to the transducer. When the sacral plexus was clearly visualized the image was frozen again and Time 2 was marked. The total time required to complete the visualization of the sacral plexus was calculated as Time 2 minus Time 1.

The diameter of the SP is measured in all patients in a transverse section at the notional intersection of the SP and a vertical line extending from the medial border of the obturator internus muscle. The measurement is taken by placing the caliper on the outer edge of hyperechoic epineurium. The same procedure is then repeated on the contralateral side.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pelvic pain scheduled for TVS

Exclusion Criteria:

* 18 years
* Women who have never been sexually active
* (suspected) Pelvic malignancy for example gynecological, intestinal or urological malignancy
* Premenarche
* Pregnancy
* Patients refusal to participate to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are consecutive patients of the Gynecology and Endometriosis Ambulance of the participating centres.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of scans to gain competency for the visualization of sacral nerve roots and sacral plexus on gynecological transvaginal ultrasound | 12 months
  The LC-CUSUM test will be used to monitor the performance of sequential interventions. Hereby the Null hypothesis (H0, performance is inadequate) is continuously tested against the alternative hypothesis (H1, performance is adequate). Negative scores for correct interventions and positive scores for incorrect results are calculated as previously reported by Biau et al. (2008a,b). Once the summation score reaches a predefined level (h) the test rejects the null hypothesis in favour of the alternative hypothesis indicating that the performance is adequate. After the literature(Tammaa 2014 and Ong 2020) we have chosen h: 1.25, P0: 0.175 as an unacceptable failure rate, and P1: 0.1, as an acceptable failure rate.

SECONDARY OUTCOMES:
inter and intraobserver variability | 12 months
  The LC-CUSUM test will be used to monitor the performance of sequential interventions. Hereby the Null hypothesis (H0, performance is inadequate) is continuously tested against the alternative hypothesis (H1, performance is adequate). Negative scores for correct interventions and positive scores for incorrect results are calculated as previously reported by Biau et al. (2008a,b). Once the summation score reaches a predefined level (h) the test rejects the null hypothesis in favour of the alternative hypothesis indicating that the performance is adequate. After the literature(Tammaa 2014 and Ong 2020) we have chosen h: 1.25, P0: 0.175 as an unacceptable failure rate, and P1: 0.1, as an acceptable failure rate
differences between sonographers of different level of experience in the field of gynecological TVS. | 12 months
  The LC-CUSUM test will be used to monitor the performance of sequential interventions. Hereby the Null hypothesis (H0, performance is inadequate) is continuously tested against the alternative hypothesis (H1, performance is adequate). Negative scores for correct interventions and positive scores for incorrect results are calculated as previously reported by Biau et al. (2008a,b). Once the summation score reaches a predefined level (h) the test rejects the null hypothesis in favour of the alternative hypothesis indicating that the performance is adequate. After the literature(Tammaa 2014 and Ong 2020) we have chosen h: 1.25, P0: 0.175 as an unacceptable failure rate, and P1: 0.1, as an acceptable failure rate
differences between participating centers. | 12 months
  The LC-CUSUM test will be used to monitor the performance of sequential interventions. Hereby the Null hypothesis (H0, performance is inadequate) is continuously tested against the alternative hypothesis (H1, performance is adequate). Negative scores for correct interventions and positive scores for incorrect results are calculated as previously reported by Biau et al. (2008a,b). Once the summation score reaches a predefined level (h) the test rejects the null hypothesis in favour of the alternative hypothesis indicating that the performance is adequate. After the literature(Tammaa 2014 and Ong 2020) we have chosen h: 1.25, P0: 0.175 as an unacceptable failure rate, and P1: 0.1, as an acceptable failure rate

CONTACTS AND LOCATIONS:
Overall Officials: Gábor Szabó, PhD, Principal Investigator — Semmelweis University
Locations (1):
- Gábor Szabó, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Szabo G, Madar I, Hudelist G, Aranyi Z, Turtoczki K, Rigo J Jr, Acs N, Liptak L, Fancsovits V, Bokor A. Visualization of sacral nerve roots and sacral plexus on gynecological transvaginal ultrasound: feasibility study. Ultrasound Obstet Gynecol. 2023 Aug;62(2):290-299. doi: 10.1002/uog.26204. PMID 36938682
- [Result] Fischerova D, Santos G, Wong L, Yulzari V, Bennett RJ, Dundr P, Burgetova A, Barsa P, Szabo G, Sousa N, Scovazzi U, Cibula D. Imaging in gynecological disease (26): clinical and ultrasound characteristics of benign retroperitoneal pelvic peripheral-nerve-sheath tumors. Ultrasound Obstet Gynecol. 2023 Nov;62(5):727-738. doi: 10.1002/uog.26223. PMID 37058402